CLINICAL TRIAL: NCT04806698
Title: Long-term Efficacy of Orthokeratology Contact Lens Wear in Controlling the Progression of Childhood Myopia
Acronym: MCOS7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menicon Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCOS7
Record Dates: First submitted 2021-03-10; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Myopia, Progressive; Children, Only
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menicon Z Night (Experimental): The experimental arm includes a group of children wearing Menicon Z Night orthokeratology contact lenses for 7 years
  Interventions: Device: Menicon Z Night
- Control (Active Comparator): The active comparator arm includes a control group of children wearing distance, single-vision glasses or soft contact lenses
  Interventions: Device: Control

INTERVENTIONS:
Device: Menicon Z Night — Children wearing Menicon Z Night orthokeratology contact lenses
  Arms: Menicon Z Night
Device: Control — Children wearing distance single-vision glasses or distance single-vision soft contact lenses
  Arms: Control

SUMMARY:
To assess the long-term efficacy of the Menicon Z Night orthokeratology contact lens in controlling the progression of childhood myopia

DETAILED DESCRIPTION:
This prospective, controlled, parallel, longitudinal study compared the axial length growth of white European myopic children wearing Menicon Z Night orthokeratology contact lenses to a control group over a 7-year period.

ELIGIBILITY:
Inclusion Criteria:

* Be 6 to 12 years of age, both ages inclusive
* A low-to-moderate level of myopia (between -0.75 and -4.00 D) and of astigmatism (≤ 1.00 D)
* Neophyte contact lens wearer
* Be successfully fitted with spectacles or orthokeratology contact lenses
* Be able to achieve, through spherical refraction correction, a logMAR visual acuity of 0.8 or better in each eye
* Be willing and able to follow the subject instructions and to meet the protocol-specified schedule of follow-up visits
* White European ethnicity

Exclusion Criteria:

* Systemic or ocular disease affecting ocular health
* Use of any systemic or topical medications that could affect ocular physiology or contact lens performance
* Any lid or anterior segment abnormalities for which contact lens wear could be contraindicated
* CCLRU grade ≥ 2 for any given anterior segment ocular clinical signs
* Aphakic, amblyopic, and atopic individuals
* Refractive astigmatism ≥ ½ spherical refraction
* Previous contact lens wear

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — White European
Enrollment: 30 (Actual)
Dates: Start 2007-03-01 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2015-03-01 (Actual)

PRIMARY OUTCOMES:
Axial length | Seven years
  To compare the axial length growth of white European myopic children wearing Menicon Z Night orthokeratology contact lenses to a control group of distance, single vision glasses or soft contact lenses

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Santodomingo-Rubido J, Villa-Collar C, Gilmartin B, Gutierrez-Ortega R, Sugimoto K. Long-term Efficacy of Orthokeratology Contact Lens Wear in Controlling the Progression of Childhood Myopia. Curr Eye Res. 2017 May;42(5):713-720. doi: 10.1080/02713683.2016.1221979. Epub 2016 Oct 21. PMID 27767354